CLINICAL TRIAL: NCT02105896
Title: Clinical Evaluation of Total-Etch and Self-Etch Dental Adhesives - 6 Year Recall
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Dentsply International (Industry)
Responsible Party: Principal Investigator, Lee Boushell, DMD, MS, Associate Professor, Operative Dentistry, University of North Carolina, Chapel Hill
Other Study IDs: 13-2235
Record Dates: First submitted 2014-03-27; First posted 2014-04-07 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Dental Bonding
Keywords: dental bonding

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: To evaluate the performance of several dental adhesives used for bonding tooth-colored fillings to teeth 6 years after the fillings have been placed.

Participants: Subjects which had participated in the study entitled "Clinical Evaluation of New Total-Etch and Self-Etch Dental Adhesives" (IRB Study #07-0673).

Procedures (methods): Fillings that had been placed 6 years ago will be evaluated by a direct, visual examination. Close-up intra-oral clinical photographs of each filling will be made. An impression of the filling may be obtained.

The specific study aim of this 6-year recall of the patients treated in IRB Study #07-0673 is to evaluate the fillings placed according to the following characteristics: Retention; Color match; Cavosurface margin discoloration; Secondary caries; Anatomic form; Marginal adaptation and/or integrity; Post-operative sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in a 2007 study entitled "Clinical Evaluation of New Total-Etch and Self-Etch Dental Adhesives" (UNC IRB Study #07-0673).

Exclusion Criteria:

* none

Ages: 25 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who participated in a 2007 study entitled "Clinical Evaluation of New Total-Etch and Self-Etch Dental Adhesives" (UNC IRB Study #07-0673).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6-year follow-up in retention. | sole visit (6 years post participation in related study).
  Each filling will be evaluated using the same modified United States Public Health Service (USPHS) direct evaluation procedures as were used during the 07-0673 study. Intraoral clinical photos will be obtained. Polyvinylsiloxane impressions of the filling and adjacent tooth structure may be obtained for those patients who had impressions made during the 07-0673 study.

SECONDARY OUTCOMES:
Change from baseline to 6-year follow-up in color match. | sole visit (6 years post participation in related study).
  Each filling will be evaluated using the same modified United States Public Health Service (USPHS) direct evaluation procedures as were used during the 07-0673 study. Intraoral clinical photos will be obtained. Polyvinylsiloxane impressions of the filling and adjacent tooth structure may be obtained for those patients who had impressions made during the 07-0673 study.

OTHER OUTCOMES:
Change from baseline to 6-year follow-up in cavosurface margin discoloration. | sole visit (6 years post participation in related study).
  Each filling will be evaluated using the same modified United States Public Health Service (USPHS) direct evaluation procedures as were used during the 07-0673 study. Intraoral clinical photos will be obtained. Polyvinylsiloxane impressions of the filling and adjacent tooth structure may be obtained for those patients who had impressions made during the 07-0673 study.
Change from baseline to 6-year follow-up in secondary caries. | sole visit (6 years post participation in related study).
  Each filling will be evaluated using the same modified United States Public Health Service (USPHS) direct evaluation procedures as were used during the 07-0673 study. Intraoral clinical photos will be obtained. Polyvinylsiloxane impressions of the filling and adjacent tooth structure may be obtained for those patients who had impressions made during the 07-0673 study.
Change from baseline to 6-year follow-up in anatomic form. | sole visit (6 years post participation in related study).
  Each filling will be evaluated using the same modified United States Public Health Service (USPHS) direct evaluation procedures as were used during the 07-0673 study. Intraoral clinical photos will be obtained. Polyvinylsiloxane impressions of the filling and adjacent tooth structure may be obtained for those patients who had impressions made during the 07-0673 study.
Change from baseline to 6-year follow-up in marginal adaptation and/or integrity. | sole visit (6 years post participation in related study).
  Each filling will be evaluated using the same modified United States Public Health Service (USPHS) direct evaluation procedures as were used during the 07-0673 study. Intraoral clinical photos will be obtained. Polyvinylsiloxane impressions of the filling and adjacent tooth structure may be obtained for those patients who had impressions made during the 07-0673 study.
Change from baseline to 6-year follow-up in post-operative sensitivity. | sole visit (6 years post participation in related study).
  Each filling will be evaluated using the same modified United States Public Health Service (USPHS) direct evaluation procedures as were used during the 07-0673 study. Intraoral clinical photos will be obtained. Polyvinylsiloxane impressions of the filling and adjacent tooth structure may be obtained for those patients who had impressions made during the 07-0673 study.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Boushell, DMD, MS, Principal Investigator — The University of North Carolina School of Dentistry
Locations (1):
- The University of North Carolina School of Dentistry, Chapel Hill, North Carolina, United States